CLINICAL TRIAL: NCT01335347
Title: A Dose Escalation Phase 1 Safety and Immunogenicity Study of an Oral Viral Vector Vaccine Encoding Avian Influenza H5N1 Hemagglutinin Protein and dsRNA Adjuvant in Healthy Adults
Brief Title: Safety Study of an Oral Vaccine to Prevent Avian Influenza
Acronym: H5N1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VXA01-001
Record Dates: First submitted 2011-04-10; First posted 2011-04-14 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Avian Influenza; Bird Flu
Keywords: Influenza; pandemic; avian influenza; H5N1; flu
MeSH Terms: conditions — Influenza in Birds; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental Low Dose (Experimental): Biological: One dose of a live replication incompetent adenovirus given in a capsule
  Interventions: Biological: ND1.1
- Experimental Medium Dose (Experimental): Biological: One or two doses of replication incompetent adenovirus given in a capsule
  Other: Placebo capsules of the same size and shape
  Interventions: Biological: ND1.1
- Experimental High Dose (Experimental): Biological: One dose of replication incompetent adenovirus in a capsule
  Interventions: Biological: ND1.1
- Placebo Control (Placebo Comparator): Capsules of the same size and shape as the experimental
  Interventions: Biological: Placebo control

INTERVENTIONS:
Biological: ND1.1 — adenovirus with the dsRNA adjuvant, dried and put into capsules
  Other Names: Ad-HA-dsRNA
  Arms: Experimental High Dose; Experimental Low Dose; Experimental Medium Dose
Biological: Placebo control — Capsules of the same size and shape as experimental groups
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to demonstrate the safety and immunogenicity of an oral vaccine to prevent avian influenza. Volunteers will receive either one or two doses of research vaccine or placebo as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* In good health as established by medical history, physical examination and laboratory testing at the time of enrollment.

Exclusion Criteria:

* Has had any other vaccines within the past 8 weeks.
* Has had prior H5 avian influenza investigational vaccine.
* Current history of chronic alcohol consumption and/or illicit and/or recreational drug use.
* History of autoimmune related disease.
* History of any confirmed or suspected immunodeficient or immunosuppressive condition (no congenital or acquired condition that impedes normal immune response, no concurrent immunosuppressive therapy).
* Positive serology for HIV, HCV, or HBV.
* Previous serious reactions to vaccination such as anaphylaxis, respiratory problems, hives or abdominal pain.
* History of irritable bowel disease or other inflammatory digestive or gastrointestinal conditions that could affect the intended distribution or safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine.
* Use of proton pump inhibitors (Nexium, Prilosec) that substantially increases stomach pH.
* Stool sample with occult blood at baseline exam

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Frequency or severity of vaccine related events as measured through reported AEs | up to 1 year

SECONDARY OUTCOMES:
Magnitude of humoral immune responses to avian influenza as measured by functional assays | up to 1 year
Magnitude of cellular immune responses to avian influenza as measured by functional assays | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sean N Tucker, PhD, Study Director — Vaxart; Martin Kabongo, MD, PhD, Principal Investigator — Accelovance
Locations (1):
- San Diego, California, United States

REFERENCES:
- [Derived] Peters W, Brandl JR, Lindbloom JD, Martinez CJ, Scallan CD, Trager GR, Tingley DW, Kabongo ML, Tucker SN. Oral administration of an adenovirus vector encoding both an avian influenza A hemagglutinin and a TLR3 ligand induces antigen specific granzyme B and IFN-gamma T cell responses in humans. Vaccine. 2013 Mar 25;31(13):1752-8. doi: 10.1016/j.vaccine.2013.01.023. Epub 2013 Jan 25. PMID 23357198